CLINICAL TRIAL: NCT02932670
Title: Minimum Effective Volume of Lidocaine for Ultrasound-Guided Costoclavicular Infraclavicular Brachial Plexus Block
Brief Title: Minimum Effective Volume of Lidocaine Costoclavicular Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, De Tran, MD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Montreal General Hospital
Record Dates: First submitted 2016-10-12; First posted 2016-10-13 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Upper Extremity Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- costoclavicular inflaclavicular block (Active Comparator): costoclavicular block with similar volume
  Interventions: Other: costoclavicular nerve block
- costoclavicular block (Experimental): costoclavicular block with decreasing volume
  Interventions: Other: costoclavicular nerve block

INTERVENTIONS:
Other: costoclavicular nerve block — ultrasound-guided costoclavicular nerve block

SUMMARY:
The aim of this study is to determine the minimum effective volume of lidocaine in 90% of patients (ED90) required for single-injection US-guided costoclavicular infraclavicular.

DETAILED DESCRIPTION:
The aim of this study is to determine the minimum effective volume of lidocaine in 90% of patients (ED90) required for single-injection US-guided costoclavicular ICB. Determination of the minimum effective volume of LA is important because it prevents the administration of an unnecessarily large (and potentially toxic) dose. Furthermore, when multiple blocks need to be performed at the same time in the same patient, knowledge of the minimum effective volume allows to the operator to preserve efficacy without sacrificing safety for each block.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 70 years
* American Society of Anesthesiologists classification 1-3
* body mass index between 20 and 30

Exclusion Criteria:

* adults who are unable to give their own consent
* pre-existing neuropathy (assessed by history and physical examination)
* coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. platelets≤ 100, International Normalized Ratio≥ 1.4 or partial prothrombin time ≥ 50)
* renal failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. creatinine≥ 100)
* hepatic failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. transaminases≥ 100)
* allergy to local anesthetics
* pregnancy
* prior surgery in the infraclavicular region
* chronic pain syndromes requiring opioid intake at home

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10; Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
success rate | 0-30 min
  minimal composite score of 14 out of 16

CONTACTS AND LOCATIONS:
Overall Officials: De QH Tran, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sotthisopha T, Elgueta MF, Samerchua A, Leurcharusmee P, Tiyaprasertkul W, Gordon A, Finlayson RJ, Tran DQ. Minimum Effective Volume of Lidocaine for Ultrasound-Guided Costoclavicular Block. Reg Anesth Pain Med. 2017 Sep/Oct;42(5):571-574. doi: 10.1097/AAP.0000000000000629. PMID 28723837